CLINICAL TRIAL: NCT01674985
Title: Microtransplantation With Decitabine and Cytarabine Improves Patient Outcomes in Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Collaborators: The Second Artillery General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST/MDS-307PLAH-ASH
Record Dates: First submitted 2012-08-25; First posted 2012-08-29 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: Decitabine; microtransplantation; myelodysplastic syndromes; chemotherapy
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine and cytarabine (Experimental): induction therapy：decitabine 25mg/m2 daily for 4 days with cytarabine 150 mg/m2 daily for 7 days consolidation：decitabine 25mg/m2 daily for 4 days with cytarabine 2g/m2 q12h for 3 days
  Interventions: Biological: Microtransplantation

INTERVENTIONS:
Biological: Microtransplantation — Infusion of G-CSF mobilized HLA-mismatched peripheral blood stem cells (G-PBSC)

SUMMARY:
The purpose of this study is to investigate whether infusion of G-CSF mobilized HLA-mismatched peripheral blood stem cells (G-PBSC) combining decitabine and cytarabine chemotherapy can improve outcomes in myelodysplastic syndromes (MDS) patients.

ELIGIBILITY:
Inclusion Criteria:

* patients 10 to 90 years old with primary or treatment-related MDS or chronic myelomonocytic leukemia;
* International Prognostic Scoring System(IPSS) intermediate-1,intermediate-2,or high risk;
* bone marrow blasts > 11% or <= 10% and poor cytogenetics;
* lack of an HLA-identical donor;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* adequate cardiac and hepatorenal functions.

Exclusion Criteria:

* have an HLA-identical donor

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2013-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
complete remission | six months

SECONDARY OUTCOMES:
disease-free survival | three years

OTHER OUTCOMES:
overall survival | three years

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Hui Ai, M.D, Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Guo M, Hu KX, Yu CL, Sun QY, Qiao JH, Wang DH, Liu GX, Sun WJ, Wei L, Sun XD, Huang YJ, Qiao JX, Dong Z, Ai HS. Infusion of HLA-mismatched peripheral blood stem cells improves the outcome of chemotherapy for acute myeloid leukemia in elderly patients. Blood. 2011 Jan 20;117(3):936-41. doi: 10.1182/blood-2010-06-288506. Epub 2010 Oct 21. PMID 20966170